CLINICAL TRIAL: NCT01660568
Title: Gemcitabine in Pretreated/Refractory NK/T Cell Lymphoma
Brief Title: Gemcitabine in NK/T Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-07-043
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2012-08

CONDITIONS: NK/T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- relapsed or refractory NK/T cell lymphoma with gemcitabine

SUMMARY:
We retrospectively review patients with refractory or relapsed ENKL who received a gemcitabine-containing regimen

ELIGIBILITY:
Inclusion Criteria:

* NK/T cell lymphoma
* relapse or refractory disease
* gemcitabine containing treatment

Exclusion Criteria:

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: relapsed or refractory NK/T cell lymphoma treated with gemcitabine conatining treatment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 2012-May

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea